CLINICAL TRIAL: NCT00510367
Title: Multimodality Treatment of Primary Breast Cancer Occurring Concomitant With Pregnancy
Brief Title: Primary Breast Cancer Occurring Concomitant With Pregnancy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID01-193; NCI-2012-01578 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-07-31; First posted 2007-08-02 (Estimated); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer; Pregnancy
Keywords: Breast Cancer; FAC; Doxorubicin; Adriamycin; Rubex; 5-Fluorouracil; 5-FU; Adrucil; Efudex; Cyclophosphamide; Cytoxan; Neosar; Pregnancy
MeSH Terms: conditions — Breast Neoplasms | interventions — Fluorouracil; Cyclophosphamide; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Multimodality Treatment (Experimental): Multimodality (chemotherapy, surgery and radiation therapy) treatment:
  5-Fluorouracil + Doxorubicin + Cyclophosphamide (FAC)
  Interventions: Drug: 5-Fluorouracil; Drug: Cyclophosphamide; Drug: Doxorubicin

INTERVENTIONS:
Drug: 5-Fluorouracil — 500 mg/m^2 By Vein Daily x 2 Days
  Other Names: 5-FU; Adrucil; Efudex
Drug: Cyclophosphamide — 500 mg/m^2 By Vein On Day 1
  Other Names: Cytoxan; Neosar
Drug: Doxorubicin — 50 mg/m^2 By Vein Over 72 Hours
  Other Names: AD; Hydroxydaunomycin hydrochloride; Adriamycin; Rubex

SUMMARY:
The goal of this clinical research study is to learn the results of multimodality (chemotherapy, surgery and radiation therapy) treatment of primary breast cancer that occurs at the same time as pregnancy. Researchers want to evaluate the outcome of labor and delivery as well as evaluate the long-term health outcomes of children exposed to chemotherapy while in their mother's womb.

DETAILED DESCRIPTION:
Patients in this study will be evaluated by the Department of Breast Medical Oncology attending physician and the obstetrician. Patients who do not have an obstetrician will be referred to an obstetrician or Maternal-Fetal Medicine specialist for evaluation.

Counseling about primary breast cancer risks, staging evaluation, and breast cancer management will be provided by members of the Department of Breast Medical Oncology. Counseling about fetal health risks will be provided by the medical oncologists and the obstetrician or the Maternal-Fetal Medicine Specialist. Counseling about surgical risks will be provided by the Breast Surgical Service. Evaluation will include a medical history and physical exam. Doctors will be evaluating patients especially for the presence of metastatic disease. The date of the last menstrual period and estimated date of delivery will be recorded.

Patients in this study will have a chest radiograph with appropriate fetal shielding. Patients will have an ultrasound of the abdomen to evaluate the presence or absence of metastatic disease in the liver. If suspicious abnormalities are found, a MRI of the abdomen will be done. Scanning MRI of the thoracic spine will be performed to screen for bone metastases. Patients will have standard blood tests and a mammogram or ultrasound of the affected breast and lymph node bearing areas. Patients will have a tissue biopsy to confirm the status of the cancer. An ultrasound will also be performed to learn the age and development of the fetus.

Patients with operable primary breast cancer tumors will have surgical evaluation for surgical therapy with modified radical mastectomy or segmental mastectomy with lymph node dissection.

Patients with locally advanced breast cancers will receive systemic multi-agent chemotherapy in the presurgical setting.

Patients will have physical exams, mammograms, and ultrasounds repeated to evaluate tumor response to treatment. All patients who will receive chemotherapy will be offered systemic chemotherapy with 5-fluorouracil, doxorubicin, and cyclophosphamide (FAC).

Patients will be followed 6-12 months using the American Society of Clinical Oncology Guidelines and the Surveillance Committee Guidelines. All children will be followed until their adulthood. If the disease gets worse, patients will be treated off the study with individualized therapy. Premedication will be provided for all patients in order to decrease the risks of nausea and vomiting. When needed, adjustment in dosage of chemotherapy or modification in the way the medicines are given will be made in order to decrease any side effects.

This is an investigational study. The FDA has approved the study drugs. Their use together in this study is experimental. At least 100 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

· All patients with primary breast cancer occurring during pregnancy will be eligible for enrollment.

Exclusion Criteria:

* Patients presenting with systemic metastases at time of diagnosis.
* Patients unwilling or unable to give informed consent.
* Patients who have received radiation therapy while pregnant
* Patients who have received chemotherapy during the first trimester of pregnancy or chemotherapy other than FAC.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2001-08-07 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-07-08 (Actual)

PRIMARY OUTCOMES:
Response of Multimodality (Chemotherapy, Surgery and Radiation Therapy) Treatment of Primary Breast Cancer in Pregnant Participants | 4 months
  Ultrasound obtained after four cycles of neoadjuvant chemotherapy to assess response.

SECONDARY OUTCOMES:
Outcome of Children Exposed to Chemotherapy While in Their Mother's Womb | Health assessments performed until child reaches the age of 18.
  Health outcomes of children exposed to chemotherapy in utero documented by survey.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Litton, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Murthy RK, Theriault RL, Barnett CM, Hodge S, Ramirez MM, Milbourne A, Rimes SA, Hortobagyi GN, Valero V, Litton JK. Outcomes of children exposed in utero to chemotherapy for breast cancer. Breast Cancer Res. 2014 Dec 30;16(6):500. doi: 10.1186/s13058-014-0500-0. PMID 25547133
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org